CLINICAL TRIAL: NCT00722137
Title: A Randomized, Open-Label, Multicenter Phase 3 Study of the Combination of Rituximab, Cyclophosphamide, Doxorubicin, VELCADE, and Prednisone (VcR-CAP) or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Patients With Newly Diagnosed Mantle Cell Lymphoma Who Are Not Eligible for a Bone Marrow Transplant
Brief Title: Study of the Combination of Rituximab, Cyclophosphamide, Doxorubicin, VELCADE, and Prednisone or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-LYM-3002; 26866138-LYM-3002CTIL (Other: Israel); 2007-005669-37 (EudraCT Number); 0970313683 (Registry Identifier: TCTIN); U1111-1195-3827 (Other: WHO)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Bortezomib; Prednisone; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- R-CHOP (Active Comparator): Rituximab 375 mg/m^2, Cyclophosphamide 750 mg/m^2, Doxorubicin 50 mg/m^2, Vincristine 1.4 mg/m^2, and Prednisone 100 mg/m^2
  Interventions: Drug: Rituximab 375 mg/m^2; Drug: Cyclophosphamide 750 mg/m^2; Drug: Doxorubicin 50 mg/m^2; Drug: Prednisone 100 mg/m^2; Drug: Vincristine 1.4 mg/m^2
- VcR-CAP (Experimental): Rituximab 375 mg/m^2, Cyclophosphamide 750 mg/m^2, Doxorubicin 50 mg/m^2, VELCADE 1.3 mg/m^2, and Prednisone 100 mg/m^2
  Interventions: Drug: Rituximab 375 mg/m^2; Drug: Cyclophosphamide 750 mg/m^2; Drug: Doxorubicin 50 mg/m^2; Drug: VELCADE 1.3 mg/m^2; Drug: Prednisone 100 mg/m^2

INTERVENTIONS:
Drug: Rituximab 375 mg/m^2 — Intravenous rituximab 375 mg/m^2 on Day 1 of a 21-day (3 week) cycle for 6 cycles.
Drug: Cyclophosphamide 750 mg/m^2 — Intravenous cyclophosphamide 750 mg/m^2 on Day 1 of a 21-day (3 week) cycle for 6 cycles
Drug: Doxorubicin 50 mg/m^2 — Intravenous doxorubicin 50 mg/m^2 on Day 1 of a 21-day (3 week) cycle for 6 cycles
Drug: VELCADE 1.3 mg/m^2 — Intravenous VELCADE 1.3 mg/m^2 on Days 1,4,8, and 11of a 21-day (3 week) cycle for 6 cycles
  Arms: VcR-CAP
Drug: Prednisone 100 mg/m^2 — Oral prednisone 100 mg/m^2 on Day 1 to Day 5 of a 21-day (3 week) cycle for 6 cycles
Drug: Vincristine 1.4 mg/m^2 — Intravenous vincristine 1.4 mg/m^2 on Day 1of a 21-day (3 week) cycle for 6 cycles. Maximum of 2 mg. Participants could receive 8 cycles if a response was initially documented at the Cycle 6 assessment.
  Arms: R-CHOP

SUMMARY:
This is a randomized, open-label, multicenter, prospective study to compare the efficacy and safety of the combination of VcR-CAP to that of R-CHOP in participants who have newly diagnosed mantle cell lymphoma grade II, III or IV and who are ineligible to undergo bone marrow transplantation.

DETAILED DESCRIPTION:
The drug being tested in this study were combination of VcR-CAP and R-CHOP. Combination of VcR-CAP and R-CHOP is being tested to treat people who had mantle cell lymphoma (MCL).

The study enrolled 487 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups in a 1:1 ratio:

Treatment Group A (VcR-CAP) Treatment Group B (R-CHOP)

The study included a screening phase, a treatment phase, a short-term follow-up phase, and a long-term follow-up phase. The screening phase was up to 28 days (56 days for bone marrow evaluation) prior to randomization.

This multi-center trial was conducted worldwide. The total study duration from randomization of the first patient until the last progression-free survival (PFS) event required for the final analysis was expected to be approximately 42 months (24 months for enrollment and 18 months for follow-up) and survival follow-up every 12 weeks until death.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older (the patient must be at least the legal age limit to be able to give informed consent within the jurisdiction the study is taking place)
* Diagnosis of mantle cell lymphoma MCL (Stage II, III or IV) as evidenced by lymph node histology and either expression of cyclin D1 (in association with CD20 and CD5) or evidence of t(11;14) translocation, such as by cytogenetics, fluorescent in situ hybridization (FISH) or polymerase chain reaction (PCR). Patients with a diagnosis of Stage I MCL will not be permitted to enter study.

  - Paraffin embedded biopsy tissue block (preferably of lymph node origin) must be sent to the central laboratory for confirmation of MCL diagnosis prior to randomization. In China, a paraffin embedded lymph node biopsy tissue block must be sent for central confirmation of sample adequacy, prior to randomization
* At least 1 measurable site of disease
* No prior therapies for MCL
* Not eligible for bone marrow transplantation as assessed by the treating physician (e.g., age or the presence of co-morbid conditions that may have a negative impact on the tolerability to transplantation).
* Eastern Cooperative Oncology Group ECOG status ≤2
* Absolute neutrophil count (ANC) ≥1500 cells/µL,
* Platelets ≥100,000 cells/µL or ≥75,000 cells/µL if thrombocytopenia is considered by the investigator to be secondary to MCL (e.g., due to bone marrow infiltration or sequestration from splenomegaly).
* Alanine transaminase ≤3 x upper limit of normal (ULN)
* Aspartate transaminase ≤3 x ULN
* Total bilirubin ≤1.5 x ULN,
* Calculated creatinine clearance ≥20 mL/min.
* Female patients must be post menopausal for at least 1 year (must not have had a natural menses for at least 12 months), surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) and have a negative serum βHCG or urine pregnancy test at screening. They must also be prepared to continue birth control measures for at least 6 months after terminating treatment.
* Male patients must agree to use an acceptable method of contraception (for themselves or female partners as listed above) for the duration of the study.
* All patients (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* In order to participate in the pharmacogenomics component of this study, patients (or their legally acceptable representative) must have signed the informed consent form for pharmacogenomics research indicating willingness to participate in the pharmacogenomics component of the study. Acquisition of tumor sample collections is required for all patients (where available); all other sample collections are optional

Exclusion Criteria:

* Prior treatment with VELCADE
* Prior antineoplastic (including unconjugated therapeutic antibodies), experimental or radiation therapy, radioimmunoconjugates or toxin immunoconjugates for the treatment of MCL. In the event that a patient has received doxorubicin for the treatment of any condition, other than MCL, the maximum dose and exposure received prior to entry into this study should not exceed 150 mg/m2.

  - short course (maximum of 10 days, not exceeding 100 mg/day) prednisone or equivalent steroids are allowed to treat symptoms in patients with advanced disease who enter the screening phase and are waiting to be randomized.
* Major surgery (at the discretion of the treating physician and in consultation with the sponsor's medical monitor) within 2 weeks before randomization
* Peripheral neuropathy or neuropathic pain of Grade 2 or worse (as per the investigators assessment)
* Diagnosed or treated for a malignancy other than MCL within 1 year of randomization, or who were previously diagnosed with a malignancy other than MCL and have any radiographic or biochemical marker evidence of malignancy. Patients with completely resected basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy are not excluded.
* Active systemic infection requiring treatment and patients with known diagnosis of human immunodeficiency virus HIV or active hepatitis B (carriers of hepatitis B are permitted to enter study)
* History of allergic reaction attributable to compounds containing boron, mannitol, or hydroxybenzoates
* Known anaphylaxis or immunoglobulin E (IgE)-mediated hypersensitivity to murine proteins or to any component of rituximab including polysorbate 80 and sodium citrate dihydrate
* Female or male patients of child-bearing potential who will not use adequate contraception during the course of the study.
* Serious medical (e.g., pericardial disease, cardiac failure [New York Heart Association; NYHA Class III or IV, Attachment 12 or left ventricular ejection fraction; LVEF <50%], active peptic ulceration, uncontrolled diabetes mellitus, or acute diffuse infiltrative pulmonary disease), or psychiatric illness likely to interfere with participation in this clinical study
* Concurrent treatment with another investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2017-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (150):
- United States (9):
  - St. Francis Hosptial and Medical Center, Hartford, Connecticut
  - Center for Cancer Care at Goshen Hospital, Goshen, Indiana
  - Sinai Hospital, Baltimore, Maryland
  - Capitol Comp. Cancer Center, Jefferson City, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Legacy Pharma Research, Bismarck, North Dakota
  - Division of Hematology and Oncology Vanderbilt University, Nashville, Tennessee
  - Cancer Outreach Associates, PC, Abingdon, Virginia
- Austria (2):
  - St.Johanns Spital/Landeskrankenhaus Salzburg, Salzburg
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Belgium (9):
  - AZ Stuivenberg Oncologie/ Hematologie, Antwerp
  - AZ St Jan AV, Bruges
  - UZ Brussel Department Medical Oncology, Brussels
  - UZA Hematologie, 1e verdiep, Edegem
  - Universitair Ziekenhuis Gent - UZ GENT, Hematologie, 9K12IE 9de verdiep- polikliniek Hematologie, Ghent
  - UZ Leuven Gasthuisberg Hematologie, Leuven
  - C.H.R. Citadelle, Liège
  - Centre Hospitalier Universitaire, Liège
  - Ucl de Mont-Godinne, Yvoir
- Brazil (11):
  - Centro de Hematologia E Hemoterapia - Unicamp, Campinas
  - Fundacao Hospital Amaral Carvalho, Jaú
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Hospital Sao Lucas Puc-Rs, Porto Alegre
  - Inca - Instituto Nacional Do Cancêr, Rio de Janeiro
  - Centro de Estudos de Hematologia E Oncologia Da Fmabc, São Paulo
  - Fundacao Pio XII - Hospital de Cancer de Barretos, São Paulo
  - Hospital Ac Camargo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
  - Santa Casa de Misericórida de São Paulo, São Paulo
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
- Chile (3):
  - Hospital Clinico Universidad Catolica de Chile, Santiago
  - Hospital Del Salvador, Santiago
  - Instituto Nacional Del Cancer, Santiago
- China (9):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang University First Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Cancer Institute & Cancer Hospital, CAMS&PUMC, Beijing
  - Peking University Third Hospital, Beijing
  - Cancer hospital, Fudan University, Shanghai
  - Ruijin Hospital, Shanghai
  - Tianjin Medical University Cancer Hospital and Institute, Tianjin
- Colombia (3):
  - Clinica Reina Sofia, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
  - Hospital Universitario San Vicente de Paul, Medellín
- Czechia (3):
  - Interni hematoonkoligicka klinika, Brno
  - Interni klinika - Oddeleni klin. hematologie Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Oddeleni klinicke hematologie, Fakultni nemocnice Kralovske Vinohrady, Prague
- Germany (9):
  - Vivantes Klinikum Neukölln Klinik für Innere Medizin Hämatologie und Onkologie, Berlin
  - Vivantes Klinikum Spandau Klinik für Innere Medizin - Hämatologie, Onkologie und Gastroenterologie, Berlin
  - Städt. Kliniken Frankfurt-Hoechst Med. Klinik II - Hämatologie und Onkologie, Frankfurt
  - Tumorklinik SANAFONTIS Alpine GmbH, Freiburg im Breisgau
  - Wilhelm-Anton-Hospital Goch gGmbH Klinik für Hämatologie und internistische Onkologie, Goch
  - Klinikum Lippe-Lemgo Med. Klinik II - Hämatologie und Onkologie, Lemgo
  - Johannes-Gutenberg-Universität Mainz III. Med. Klinik, Mainz
  - Mutterhaus der Borromäerinnen Med. Klinik I, Trier
  - Schwarzwald-Baar-Kliniken Innere Med. II, Villingen
- Hungary (3):
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, III. sz. Belgyogyaszati Klinika, Debrecen
  - Petz Aladár Kórház, II. Belgyógyászat, Győr
  - Kaposi Mor Megyei Korhaz, Belgyogyaszat, Kaposvár
- India (7):
  - Apollo Hospital and Research Foundation, Apollo Hospitals, Hyderabad 500033, Andhra Pradesh
  - Kidwai Memorial Institute of Oncology, Bangalore 560 029, Karnataka
  - Regional Cancer Centre, Medical Oncology, Thiruvananthapuram, Kerala-695011
  - Jehangir Hospital, Pune-411002, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi- 110060, National Capital Territory of Delhi
  - Apollo Speciality Hospital, Chennai, Chennai-600035, Tamil Nadu
  - Netaji Subash Chanda Bose Cancer Research Institute, Kolkata- 700016, West Bengal
- Israel (5):
  - Rambam Medical Center-Hematology department, Haifa
  - Hadassah Medical Center - Hematology department, Jerusalem
  - Rabin Medical Center, Beilinson Campus, Petach Tiqva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center - Hematology Institute, Rehovot
- Italy (5):
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S.Orsola-Malpighi Dipartimento di Ematologia e Scienze Oncologiche "L. e A. Seragnoli", Bologna
  - Spedali Civili di Brescia, Brescia
  - Dipartimento di Oncologia ed Ematologia Università di Modena e Reggio Emilia, Modena
  - AZIENDA OSPEDALIERA UNIVERSITARIA POLICLINICO TOR VERGATA DIPARTIMENTO DI MEDICINA U.O.C. Ematologia, Roma
  - Azienda Ospedaliera San Giovanni Battista "Molinette" Struttura Complessa Ematologia 2, Torino
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Gleneagles Medical Centre, Pulau Pinang
- Morocco (3):
  - Hopital Du 20 Aout 1953, Casablanca
  - Centre D'oncologie Al Azhar, Rabat
  - Institut National D'oncologie, Rabat
- Philippines (2):
  - National Kidney and Transplant Institute, Quezon City
  - St Lukes Medical Center, Quezon City
- Poland (4):
  - Szpital Morski im. PCK w Gdyni Gdynskie Centrum Onkologii Oddzial Chemioterapii, Gdynia
  - Klinika Hematologii Uniwersytetu Medycznego w Lodzi, Lodz
  - "Katedra i Klinika Hematologii i Chorob Rozrostowych Ukladu Krwiotworczego, Poznan
  - Klinika Hematologii Nowotworow Krwi i Transplantacji Szpiku Akademii Medycznej we Wroclawiu, Wroclaw
- Portugal (4):
  - Hospital Sao Marcos, Braga
  - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia, Porto
- Romania (5):
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris", Hematologie, Baia Mare
  - Institutul Clinic Fundeni, Hematologie, Bucharest
  - Spitalul Clinic Coltea, Clinica Hematologie, Bucharest
  - Spitalul Clinic Universitar de Urgenta Bucuresti, Hematologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta "Sf. Spiridon" Iasi, Oncologie Medicala, Iași
- Russia (20):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Belgorod Regional Oncology Center, Belgorod
  - Chelyabinsk Regional Oncology Center, Chelyabinsk
  - 1st Republican Clinical Hospital of Udmurtia, Izhevsk
  - Cancer Research Center RAMS - N.N. Blokhin - Academy of Medical Science, Moscow
  - Hematology Scientific Center, Moscow
  - Moscow Regional Clinical Research Institute, Moscow
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Medical Scientific Radiology - Center, Obninsk
  - Omsk Regional Oncology Dispensary, Omsk
  - Medical Sanitary Unit # 1, Perm
  - Republikan Hospital named after V.A/ Baranov, Petrozavodsk
  - Rostov Research Institute of Oncology, Rostov-on-Don
  - Central Res. Inst. of Roentgen-Radiology, Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Leningrad Region Clinical Hospital, Saint Petersburg
  - Pavlov State Medical Univercity, Saint Petersburg
  - St.-Petersburg Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Sverdlovsk Regional Oncology Dispensary, Yekaterinburg
- Singapore (2):
  - National Cancer Centre, Singapore
  - Singapore General Hospital - Hematology, Singapore
- South Africa (5):
  - Chris Hani Baragwanath Hospital, Johannesburg, Gauteng
  - Medical Oncology Center of Rosebank, Johannesburg, Gauteng
  - University of the Witwatersrand Oncology, Johannesburg, Gauteng
  - Pretoria Academic Hospital-Dr. Savage Road, 3rd Floor Radiotherapy Building, Prinshof, Pretoria, Gauteng
  - Dr AI Pirjol & Dr WM Szpak Inc., Durban, KwaZulu-Natal
- Spain (5):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital de la Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Salamanca, Salamanca
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital-Hematology Unit, Bangkok
  - Maharaj Nakorn Chiang Mai hospital - Faculty of Medicine, Chiang Mai
- Tunisia (4):
  - Hôpital Farhat Hached, Sousse
  - Centre National de Greffe de Moelle osseuse, Tunis
  - Hôpital Aziza Othmana, Tunis
  - Institut Salah Azaiz, Tunis
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Dokuz Eylul University Med. Fac., Izmir
- Ukraine (7):
  - Cherkassy Regional Oncology Center, Dept. of Hematology, Cherkassy
  - Dnepropetrovsk City Clinical Hospital #4, Regional Hematology Center, Dnipro
  - Institute of Urgent and Recovery Surgery named after V.K.Gusaka of AMS of Ukraine, Haematology Dept., Donetsk
  - Khmelnitskiy Regional Hospital, Hematology Department, Khmelnitsky
  - National Cancer Institute, Department of chemotherapy of hemoblastosis, Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Lviv Clinical Hospital #5, Hematology Dept., Lviv
  - Crimean Republic Clinical Oncology Dispensary, Haematology Department, Simferopol

REFERENCES:
- [Derived] Robak T, Jin J, Pylypenko H, Verhoef G, Siritanaratkul N, Drach J, Raderer M, Mayer J, Pereira J, Tumyan G, Okamoto R, Nakahara S, Hu P, Appiani C, Nemat S, Cavalli F; LYM-3002 investigators. Frontline bortezomib, rituximab, cyclophosphamide, doxorubicin, and prednisone (VR-CAP) versus rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in transplantation-ineligible patients with newly diagnosed mantle cell lymphoma: final overall survival results of a randomised, open-label, phase 3 study. Lancet Oncol. 2018 Nov;19(11):1449-1458. doi: 10.1016/S1470-2045(18)30685-5. Epub 2018 Oct 19. PMID 30348538
- [Derived] Robak T, Huang H, Jin J, Zhu J, Liu T, Samoilova O, Pylypenko H, Verhoef G, Siritanaratkul N, Osmanov E, Pereira J, Mayer J, Hong X, Okamoto R, Pei L, Rooney B, van de Velde H, Cavalli F. Association between bortezomib dose intensity and overall survival in mantle cell lymphoma patients on frontline VR-CAP in the phase 3 LYM-3002 study. Leuk Lymphoma. 2019 Jan;60(1):172-179. doi: 10.1080/10428194.2017.1321750. Epub 2017 Jun 5. PMID 28583031
- [Derived] Verhoef G, Robak T, Huang H, Pylypenko H, Siritanaratkul N, Pereira J, Drach J, Mayer J, Okamoto R, Pei L, Rooney B, Cakana A, van de Velde H, Cavalli F. Association between quality of response and outcomes in patients with newly diagnosed mantle cell lymphoma receiving VR-CAP versus R-CHOP in the phase 3 LYM-3002 study. Haematologica. 2017 May;102(5):895-902. doi: 10.3324/haematol.2016.152496. Epub 2017 Feb 9. PMID 28183846
- [Derived] Robak T, Huang H, Jin J, Zhu J, Liu T, Samoilova O, Pylypenko H, Verhoef G, Siritanaratkul N, Osmanov E, Alexeeva J, Pereira J, Drach J, Mayer J, Hong X, Okamoto R, Pei L, Rooney B, van de Velde H, Cavalli F; LYM-3002 Investigators. Bortezomib-based therapy for newly diagnosed mantle-cell lymphoma. N Engl J Med. 2015 Mar 5;372(10):944-53. doi: 10.1056/NEJMoa1412096. PMID 25738670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 487 participants were randomized from 128 centers in 28 countries from 22 May 2008 to 17 June 2017; 244 to the R-CHOP treatment group and 243 to the VcR-CAP treatment group. Of the 487 randomized participants, 242 in the R-CHOP group and 240 in the VcR-CAP group received at least 1 dose of study drug.
Groups:
- R-CHOP: Rituximab 375 mg/m^2, Cyclophosphamide 750 mg/m^2, Doxorubicin 50 mg/m^2, Vincristine 1.4 mg/m^2 and Prednisone 100 mg/m^2 Rituximab: Rituximab intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles. Cyclophosphamide: Cyclophosphamide intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles Doxorubicin: Intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles Prednisone: Prednisone orally on Day 1 to Day 5 of a 21 day (3 week) cycle for 6 cycles Vincristine: Vincristine intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles.
- VcR-CAP: Rituximab 375 mg/m^2, Cyclophosphamide 750 mg/m^2, Doxorubicin 50 mg/m^2, VELCADE 1.3 mg/m^2, and Prednisone 100 mg/m^2 Rituximab: Rituximab intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles. Cyclophosphamide: Cyclophosphamide intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles Doxorubicin: Intravenous on Day of a 21 day (3 week) cycle for 6 cycles VELCADE: VELCADE intravenous on Days 1,4,8, and 11 of a 21 day (3 week) cycle for 6 cycles Prednisone: Prednisone orally on Day 1 to Day 5 of a 21 day (3 week) cycle for 6 cycles.
Period: Overall Study
Arm/Group | R-CHOP | VcR-CAP
Started | 244 | 243
Completed (Completed participants are the participants who completed the treatment.) | 199 | 195
Not Completed | 45 | 48
Not completed — Overt Disease Progression | 5 | 4
Not completed — Adverse Event | 17 | 21
Not completed — Death | 12 | 7
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Other Reason Unknown | 3 | 4
Not completed — Randomized But Not Treated | 2 | 3

BASELINE CHARACTERISTICS:
Population: The population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | R-CHOP | VcR-CAP | Total
Number analyzed (Participants) | 244 | 243 | 487
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.78) | 64.2 (9.68) | 64.3 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 127
  Male | 182 | 178 | 360
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 68 | 88 | 156
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 172 | 151 | 323
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 10 | 16 | 26
  Poland | 9 | 10 | 19
  Czech Republic | 5 | 9 | 14
  Spain | 8 | 6 | 14
  Hungary | 5 | 8 | 13
  Romania | 9 | 4 | 13
  Austria | 6 | 4 | 10
  Italy | 6 | 3 | 9
  Germany | 7 | 1 | 8
  Portugal | 3 | 4 | 7
  France | 1 | 2 | 3
  Canada | 6 | 1 | 7
  United States | 2 | 5 | 7
  Russia | 57 | 42 | 99
  China | 34 | 61 | 95
  Ukraine | 18 | 16 | 34
  Brazil | 9 | 13 | 22
  Thailand | 9 | 10 | 19
  Japan | 11 | 7 | 18
  India | 9 | 3 | 12
  Israel | 5 | 2 | 7
  Tunisia | 3 | 3 | 6
  Turkey | 5 | 1 | 6
  Colombia | 2 | 3 | 5
  Korea, Republic Of | 2 | 3 | 5
  Chile | 1 | 2 | 3
  Singapore | 1 | 2 | 3
  Taiwan, Province Of China | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the interval between the date of randomization and the date of progressive disease (PD) or death, whichever occurred first. PD was based on the assessment of an Independent Review Committee.
Time Frame: Median duration of follow-up of 40 months
Population: The population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 244 | 243
Days | 437.0 [365.0 to 513.0] | 751.0 [604.0 to 969.0]
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p < 0.001, Log Rank; Based on Log rank test stratified with International Prognostic Index (IPI) risk and stage of disease; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.50 to 0.79] — Hazards ratio estimate is based on a Cox´s model stratified by IPI risk and stage of disease. A hazard ratio < 1 indicates an advantage for VcR-CAP

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression was defined as the duration from the date of randomization until the date of first documented evidence of progressive disease (PD) or date of relapse for subjects who experienced complete response (CR) or complete response, unconfirmed (CRu). PD and response were based on the assessment of an Independent Review Committee.
Time Frame: Median duration of follow-up of 40 months
Population: The population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 244 | 243
Days | 490.0 [417.0 to 550.0] | 929.0 [696.0 to 1245.0]
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p < 0.001, Log Rank; Based on Log rank test stratified with IPI risk and stage of disease; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.45 to 0.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Duration of Response
Description: The duration of treatment response was defined as the time from the date of the first response to the date of PD or death due to PD for those participants with a best response of CR, CRu, or PR as determined by the Independent Review Committee. The duration of response for complete responders was defined as the time from the date of the first response to the date of PD or death due to PD for those participants with a best response of CR or CRu verified by bone marrow and lactate dehydrogenase (LDH).
Time Frame: Median duration of follow-up of 40 months
Population: The response-evaluable population was defined as all participants who received at least 1 dose of study drug, had >= 1 measurable tumor mass (>1.5 cm in the longest dimension and >1.0 cm in the short axis) at baseline and had at least 1 post-baseline tumor assessment by Independent Review Committee, before any subsequent anti-lymphoma treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 228 | 229
Days
  Duration of response: number analyzed (Participants) | 204 | 211
  Duration of response | 459.0 [379.0 to 518.0] | 1110.0 [813.0 to 1320.0]
  Duration for Complete responders: number analyzed (Participants) | 95 | 122
  Duration for Complete responders | 563.0 [486.0 to 738.0] | 1282.0 [933.0 to 1602.0]

4. Secondary Outcome: Time to Next Anti-lymphoma Treatment (TTNT)
Description: The time to next anti-lymphomatreatment was measured from the date of initiation of study treatment as per protocol to the start date of new anti-lymphoma treatment. Death due to disease progression prior to subsequent therapy was considered as an event. Otherwise, time to next anti lymphoma treatment was censored at the date of death or the last date known to be alive.
Time Frame: : Median duration of follow-up of 40 months
Population: The population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 244 | 243
Days | 756.0 [674.0 to 837.0] | 1353.0 [1180.0 to NA] — The upper limit of the confidence interval was not able to be estimated.
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p < 0.001, Log Rank; Based on Log rank test stratified with IPI risk and stage of disease; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.38 to 0.65] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Treatment-free Interval (TFI)
Description: The TFI was defined as the duration from the date of last dose plus 1 day to the start date of the new treatment. Death due to disease progression prior to subsequent therapy was considered as an event. Otherwise, treatment-free interval was censored at the date of death or the last date known to be alive.
Time Frame: Median duration of follow-up of 40 months
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 242 | 240
Days | 624.0 [542.0 to 693.0] | 1236.0 [1023.0 to NA] — The upper limit of the confidence interval was not able to be estimated.
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.38 to 0.65]

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as complete response (CR) + complete response, unconfirmed (CRu) + partial response (PR) as determined by the Independent Review Committee. Response assessment was carried out every 6 weeks for 18 weeks; thereafter, every 8 weeks until PD/initiation of alternate therapy/withdrawal from study/death.
Time Frame: Median duration of follow-up of 40 months
Population: The response-evaluable population was defined as all participants who received >= 1 dose of study drug, had at least 1 measurable tumor mass (>1.5 cm in the longest dimension and >1.0 cm in the short axis) at baseline and had at least 1 post-baseline tumor assessment by Independent Review Committee, before any subsequent anti-lymphoma treatment.
Measure: Number; unit: Participants
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 228 | 229
Participants | 204 | 211
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p = 0.275, Cochran-Mantel-Haenszel Chi-Square; Odds Ratio (OR) = 1.428, 95% CI 2-sided [0.749 to 2.722] — Mantel-Haenszel estimate of the common odds ratio for stratified tables is used, with IPI risk and Stage of Disease as stratification factors. An odds ratio (OR) > 1 indicates an advantage for VcR-CAP

7. Secondary Outcome: Overall Complete Response (CR + CRu)
Description: Overall complete response was defined as the number of participants with complete response (CR) and those with unconfirmed complete response (CRu). Response assessment was carried out every 6 weeks for 18 weeks; thereafter, every 8 weeks until PD/initiation of alternate therapy/withdrawal from study/death.
Time Frame: Median duration of follow-up of 40 months
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 228 | 229
Participants
  Overall complete response | 95 | 122
  CR | 79 | 106
  CRu | 16 | 16
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p < 0.007, Cochran-Mantel-Haenszel Chi-Square; Odds Ratio (OR) = 1.688, 95% CI 2-sided [1.148 to 2.481] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from the date of randomization to the date of the participant's death. If the participant was alive or the vital status was unknown, OS was censored at the date that the subject was last known to be alive.
Time Frame: Median duration of follow-up of 40 months
Population: The population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 244 | 243
Days | 1714.0 [1436.0 to NA] — The upper limit of the confidence interval was not able to be estimated. | NA [1704.0 to NA] — The median was not reached and the upper limit of the confidence interval was not able to be estimated.
Statistical Analysis 1: Comparison: R-CHOP vs VcR-CAP; Test type: Superiority or Other; p = 0.173, Log Rank; Based on Log rank test stratified with IPI risk and stage of disease; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.59 to 1.10] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: 18-Month Survival
Description: 18-month survival was defined as the estimated probability of survival at 18 months (Kaplan-Meier estimate).
Time Frame: Up to month 18 from the time of randomization
Population: The population consisted of all randomized participants.
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 83.8 [78.4 to 87.9] | 84.9 [79.6 to 88.9]

10. Secondary Outcome: Overall Survival (OS) in Long Term Follow-up Period
Description: as for outcome 8
Time Frame: Up to 107.4 months
Population: The population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 244 | 243
Days | 1695.0 [1436.0 to 2098.0] | 2760.0 [2172.0 to NA] — Upper limit of overall survival after long term follow-up was not estimable due low number of participants with the event.

11. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug, whether or not considered drug related. AEs were collected from the first dose of study drug through 30 days after the last dose of study drug. Treatment was administered for up to 8 cycles (24 weeks) and AEs were collected for up to 30 days following the last dose of study drug.
Time Frame: Up to 107.4 months
Population: The safety population was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | R-CHOP | VcR-CAP
Number analyzed (Participants) | 242 | 240
Participants | 239 | 240

ADVERSE EVENTS:
Time Frame: Up to 107.4 months
Description: The safety population was defined as all randomized participants who received at least 1 dose of study medication.
Arm/Group | R-CHOP | VcR-CAP
Serious Adverse Events (participants affected / at risk) | 72/242 | 91/240
Other Adverse Events (participants affected / at risk) | 187/242 | 185/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP (N=242) | VcR-CAP (N=240)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 26
Neutropenia (Blood and lymphatic system disorders) | 13 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 8
Leukopenia (Blood and lymphatic system disorders) | 3 | 6
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 19
Sepsis (Infections and infestations) | 1 | 4
Bronchitis (Infections and infestations) | 2 | 2
Lobar pneumonia (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 1 | 2
Pneumonia streptococcal (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 1 | 2
Abscess neck (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1
Candidiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 10
Acute phase reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Cardiac death (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Periproctitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 2
Poor venous access (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 2
Autonomic neuropathy (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — This serious adverse event occurred during long term follow-up period
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP (N=242) | VcR-CAP (N=240)
Nausea (Gastrointestinal disorders) | 33 | 59
Abdominal distension (Gastrointestinal disorders) | 5 | 22
Abdominal pain (Gastrointestinal disorders) | 9 | 18
Abdominal pain upper (Gastrointestinal disorders) | 11 | 16
Dyspepsia (Gastrointestinal disorders) | 14 | 13
Neuropathy peripheral (Nervous system disorders) | 19 | 19
Paraesthesia (Nervous system disorders) | 12 | 16
Dizziness (Nervous system disorders) | 9 | 15
Hypoaesthesia (Nervous system disorders) | 15 | 15
Headache (Nervous system disorders) | 11 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 49
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 33 | 33
Rash (Skin and subcutaneous tissue disorders) | 8 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 14
Insomnia (Psychiatric disorders) | 18 | 27
Weight decreased (Investigations) | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-01-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT00722137/SAP_000.pdf
  • Study Protocol (2014-02-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT00722137/Prot_001.pdf